CLINICAL TRIAL: NCT04218877
Title: Trigger's Influence on Atopic Dermatitis Manifestation in Children Under 3 Years Old
Brief Title: The Factors Affecting Atopic Dermatitis in Children Age 1-3
Status: Completed | Type: Observational
Sponsor: Akusherstvo Pro (Other)
Responsible Party: Sponsor
Other Study IDs: AkusherstvoPro
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with atopic dermatitis: Children 1-3 years old with atopic dermatitis
- Children without atopic dermatitis
- Children with genetic predisposition: Children with genetic predisposition to atopic dermatitis, but without manifestations

INTERVENTIONS:
Other:  — There will be no intervention, only observation

SUMMARY:
This study evaluates the influence of different triggers on atopic dermatitis manifestation in children under 3 years old.

DETAILED DESCRIPTION:
In this study investigators evaluate the influence of atopic dermatitis triggers before labour, right after labour, in firsts weeks after labour, in first year. Investigators want to find the most popular and most important factors witch provoke atopic dermatitis manifestation and comparison the results with children without atopic dermatitis but with genetic predisposition to it.

ELIGIBILITY:
Inclusion Criteria:

* children 1-3 age without rash, without atopic dermatitis
* children 1-3 age with recurrent atopic dermatitis

Exclusion Criteria:

* children 1-3 age with non-specific rush
* children age 1-2 with atopic dermatitis without rush during previous year

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients A Medclinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Trigger's factors for atopic dermatitis | 3 years
  Vitamins during pregnancy; probiotics during pregnancy; school for future parents; vaginal birth; cesarian section; "golden hour" after delivery; antibiotics for mother and child right away after delivery; vaccination; breastfeeding; time after delivery for discharging hospital; using herbs for child's bathing; cosmetics for child; mother's diet after delivery; air's moisture; newborn's acne; pets; in what age child taste egg, cow's milk, fish, wheat, peanut, seafood; breastfeeding durations; infant formula in first year. All this factor will be aggregated as "yes" and "no"

CONTACTS AND LOCATIONS:
Locations (1):
- Amedclinic, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No